CLINICAL TRIAL: NCT00524745
Title: Comparison of the Immunogenicity and Reactogenicity of Alternative Schedules of Gardasil Vaccine to Prevent HPV Infection
Brief Title: Immunogenicity and Reactogenicity of Alternative Schedules of Gardasil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPV01
Record Dates: First submitted 2007-08-31; First posted 2007-09-05 (Estimated); Results first posted 2011-09-08 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2012-07

CONDITIONS: Dose Schedule Study
Keywords: Gardasil; Human Papillomavirus; HPV vaccine; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Vaccines, Synthetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0,2,6 month vaccination schedule (Active Comparator)
  Interventions: Biological: Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine
- 0,3,9 month vaccination schedule (Active Comparator)
  Interventions: Biological: Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine
- 0,6,12 month vaccination schedule (Active Comparator)
  Interventions: Biological: Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine
- 0,12,24 month vaccination schedule (Active Comparator)
  Interventions: Biological: Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine

INTERVENTIONS:
Biological: Biological: quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine — Three doses of quadrivalent HPV recombinant vaccine administered at different dosing intervals in each of four study arms.

SUMMARY:
To demonstrate that Gardasil® vaccine, when given to girls 11-13 years of age according to 1 of 3 alternative 3-dose schedules (0, 3, 9 months; 0, 6, 12 months; or 0, 12, 24 months), results in anti-HPV type 16 and anti-HPV type 18 responses 28 days post-dose 3 that are similar to those obtained when the vaccine is given on the standard 3-dose schedule of 0, 2, 6 months.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary objective:

To test the hypothesis that Gardasil® vaccine, when administered to girls 11-13 years of age according to 1 of 3 alternative 3-dose schedules (0,3,9 months; 0,6,12 months; or 0,12,24 months), results in anti-HPV 16 and anti-HPV 18 responses 28 days post-dose 3 that are similar to those obtained when the vaccine is administered on the standard 3-dose schedule of 0,2,6 months.

Secondary objectives:

1. To test the hypothesis that Gardasil® vaccine, when administered to girls 11-13 years of age according to 1 of 3 alternative 3-dose schedules (0,3,9 months; 0,6,12 months; or 0,12,24 months), results in anti-HPV 6 and anti-HPV 11 responses 28 days post-dose 3 that are similar to those obtained when the vaccine is administered on the standard 3-dose schedule of 0,2,6 months.
2. To describe the safety profile of the administration of Gardasil® according to each of the four schedules by assessing:

   (i) immediate reactogenicity (reactions within 30 minutes after each injection); (ii) solicited (local reactogenicity and fever) and unsolicited events occurring during the first 7 days following each vaccination; (iii) serious adverse events occurring up to one month following the last dose of vaccine; (iv) deaths or adverse events occurring at any time determined to be vaccination-related.

ELIGIBILITY:
Inclusion Criteria:

1. 11-13 years of age.
2. Signed informed consent form (both parent's & daughter's signature).
3. Good health status.
4. Able to comply with trial protocol.
5. Plans to stay at current school for duration of study.

Exclusion Criteria:

1. Prior HPV vaccination
2. Pregnant or lactating or intends to become pregnant during study period.
3. Apparent moderate or severe acute illness.
4. Clinical history of bleeding disorder such as hemophilia, thrombocytopenia, or anticoagulant therapy.
5. Clinical history of impaired immune responsiveness, whether due to use of immunosuppressive therapy, a genetic defect, HIV infection, or other causes.
6. Hypersensitivity to the active substances or to any of the excipients of the HPV vaccine, or such reactions to other vaccines received in the past.
7. Investigational drug or investigational vaccine administered during the period from 30 days before to 30 days after any dose of HPV vaccine.

Ages: 11 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 903 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Neuzil, MD, MPH, Principal Investigator — PATH
Locations (1):
- National Institute of Hygiene and Epidemiology, Hanoi, Vietnam

REFERENCES:
- [Result] Neuzil KM, Canh DG, Thiem VD, Janmohamed A, Huong VM, Tang Y, Diep NT, Tsu V, LaMontagne DS. Immunogenicity and reactogenicity of alternative schedules of HPV vaccine in Vietnam: a cluster randomized noninferiority trial. JAMA. 2011 Apr 13;305(14):1424-31. doi: 10.1001/jama.2011.407. PMID 21486975
- [Derived] Widdice LE, Unger ER, Panicker G, Hoagland R, Callahan ST, Jackson LA, Berry AA, Kotloff K, Frey SE, Harrison CJ, Pahud BA, Edwards KM, Mulligan MJ, Sudman J, Bernstein DI. Antibody responses among adolescent females receiving two or three quadrivalent human papillomavirus vaccine doses at standard and prolonged intervals. Vaccine. 2018 Feb 1;36(6):881-889. doi: 10.1016/j.vaccine.2017.12.042. Epub 2018 Jan 3. PMID 29306506
- [Derived] Lamontagne DS, Thiem VD, Huong VM, Tang Y, Neuzil KM. Immunogenicity of quadrivalent HPV vaccine among girls 11 to 13 Years of age vaccinated using alternative dosing schedules: results 29 to 32 months after third dose. J Infect Dis. 2013 Oct 15;208(8):1325-34. doi: 10.1093/infdis/jit363. Epub 2013 Jul 30. PMID 23901077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 schools were (1) matched according to size, urban/rural location and ethnicity; (2) assigned to one of four groups; and (3) randomized to one of four schedules
  All girls 11-13 years of age in these schools were eligible to participate.
Period: Overall Study
Arm/Group | 0,3,9 Month Schedule | 0,6,12 Month Schedule | 0,12,24 Month Schedule | Standard (0,2,6 Month) Schedule
Started | 229 | 206 | 241 | 227
Completed | 195 | 193 | 212 | 205
Not Completed | 34 | 13 | 29 | 22
Not completed — subject withdrawal or lost to follow up | 34 | 13 | 29 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0,3,9 Month Schedule | 0,6,12 Month Schedule | 0,12,24 Month Schedule | Standard (0,2,6 Month) Schedule | Total
Number analyzed (Participants) | 229 | 206 | 241 | 227 | 903
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 229 | 206 | 241 | 227 | 903
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 206 | 241 | 227 | 903
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 229 | 206 | 241 | 227 | 903

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Antibody Response to HPV Type 16 1 Month Post-dose 3 for Each Alternative Schedule Compared to the Standard Schedule.
Time Frame: 25 months
Measure: Number (95% Confidence Interval); unit: GMT ratio
Arm/Group | 0,3,9 Month Schedule | 0,6,12 Month Schedule | 0,12,24 Month Schedule | Standard (0,2,6 Month) Schedule
Number analyzed (Participants) | 194 | 193 | 212 | 205
GMT ratio | 0.93 [0.71 to 1.21] | 0.99 [0.75 to 1.30] | 0.63 [0.48 to 0.83] | 1.0 [NA to NA] — Standard schedule is the comparator for the GMT ratio outcome reported.

2. Primary Outcome: Comparison of Antibody Response to HPV Type 18 1 Month Post-dose 3 for Each Alternative Schedule Compared to the Standard Schedule.
Time Frame: 25 months
Measure: Number (95% Confidence Interval); unit: GMT ratio
Arm/Group | 0,3,9 Month Schedule | 0,6,12 Month Schedule | 0,12,24 Month Schedule | Standard (0,2,6 Month) Schedule
Number analyzed (Participants) | 195 | 193 | 213 | 205
GMT ratio | 0.88 [0.69 to 1.12] | 0.92 [0.71 to 1.18] | 0.77 [0.62 to 0.96] | 1.0 [NA to NA] — Standard schedule is the comparator for the GMT ratio outcome reported.

3. Secondary Outcome: Comparison of Antibody Response to HPV Type 6 1 Month Post-dose 3 for Each Alternative Schedule Compared to the Standard Schedule.
Time Frame: 25 months
Measure: Number (95% Confidence Interval); unit: GMT ratio
Arm/Group | 0,3,9 Month Schedule | 0,6,12 Month Schedule | 0,12,24 Month Schedule | Standard (0,2,6 Month) Schedule
Number analyzed (Participants) | 191 | 191 | 207 | 203
GMT ratio | 1.07 [0.80 to 1.44] | 1.14 [0.85 to 1.52] | 0.64 [0.46 to 0.90] | 1.0 [NA to NA] — Standard schedule is the comparator for the GMT ratio outcome reported.

4. Secondary Outcome: Comparison of Antibody Response to HPV Type 11 1 Month Post-dose 3 for Each Alternative Schedule Compared to the Standard Schedule.
Time Frame: 25 months
Measure: Number (95% Confidence Interval); unit: GMT ratio
Arm/Group | 0,3,9 Month Schedule | 0,6,12 Month Schedule | 0,12,24 Month Schedule | Standard (0,2,6 Month) Schedule
Number analyzed (Participants) | 195 | 193 | 212 | 205
GMT ratio | 0.86 [0.70 to 1.06] | 0.86 [0.69 to 1.06] | 0.96 [0.80 to 1.15] | 1.0 [NA to NA] — Standard schedule is the comparator for the GMT ratio outcome reported.

ADVERSE EVENTS:
Time Frame: Solicited local reactions within 7 days post-vacciantion
Arm/Group | 0,3,9 Month Schedule | 0,6,12 Month Schedule | 0,12,24 Month Schedule | Standard (0,2,6 Month) Schedule
Serious Adverse Events (participants affected / at risk) | 0/229 | 0/206 | 0/241 | 0/227
Other Adverse Events (participants affected / at risk) | 157/229 | 133/206 | 148/240 | 131/227
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0,3,9 Month Schedule (N=229) | 0,6,12 Month Schedule (N=206) | 0,12,24 Month Schedule (N=240) | Standard (0,2,6 Month) Schedule (N=227)
Fever post dose 1 (General disorders) | 6 | 4 | 7 | 5 — 7-day subject diary
Fever post dose 2 (General disorders) | 5 | 2 | 4 | 6 — 7-day subject diary
Fever post-dose 3 (General disorders) | 9 | 6 | 12 | 12 — 7 day subject diary
Pain at injection site post dose 1 (General disorders) | 133 | 96 | 114 | 120 — 7 day subject diary
Pain at injection site post dose 2 (General disorders) | 124 | 124 | 134 | 117 — 7 day subject diary
Pain at injection site post dose 3 (General disorders) | 149 | 128 | 139 | 121 — 7 day subject diary

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes